CLINICAL TRIAL: NCT01859143
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of 3 New 6:2 Influenza Virus Reassortants in Adults
Brief Title: Study to Evaluate the Safety of 3 New 6:2 Influenza Virus Reassortants in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MED-VA-FLUMIST-1156
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Influenza; Healthy
Keywords: Trivalent; Influenza; FluMist Quadrivalent; Vaccine; Prevention; Healthy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trivalent Influenza Vaccine (Experimental): A single dose of 10^(7.0 +/- 0.5) fluorescent focus units (FFU) of trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Interventions: Biological: Trivalent Influenza Vaccine
- Placebo (Placebo Comparator): A single dose of placebo matched to trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine — A single dose of 10^(7.0 ± 0.5) FFU of trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Trivalent Influenza Vaccine
Other: Placebo — A single dose of placebo matched to trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Placebo

SUMMARY:
This prospective annual release study is designed to evaluate the safety on new influenza virus vaccine strains to be included in FluMist Quadrivalent for the 2013-2014 influenza season.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo-controlled release study will enroll approximately 300 healthy adults 18 to 49 years of age. Eligible subjects will be randomly assigned in a 4:1 fashion to receive a single dose of trivalent vaccine or placebo by intranasal spray. Randomization will be stratified by site. This study will be conducted at 3 sites in the United States of America. Each subject will receive 1 dose of investigational product on Day 1. The duration of study participation for each subject is the time from study vaccination through 180 days after study vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 49 years
* Written informed consent
* Subject available by telephone
* Ability to understand and comply with the requirements of the protocol, as judged by the Investigator

Exclusion Criteria:

* Concurrent enrollment in another clinical study up to 180 days after receipt of investigational product (Day 181)
* History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life threatening, or severe reactions to previous influenza vaccinations
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (example [eg], asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (greater than [>] 100.0 degrees Fahrenheit [F] oral or equivalent) and/or clinically significant respiratory illness (example, cough or sore throat) within 14 days prior to randomization
* Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Research Site, Miami, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant randomized to receive placebo received trivalent influenza vaccine on Day 1 instead of placebo and was included in trivalent influenza vaccine group in the safety population.
Groups:
- Trivalent Influenza Vaccine: A single dose of 10^(7.0 +/- 0.5) fluorescent focus units (FFU) of trivalent influenza vaccine administered as intranasal spray on Day 1.
- Placebo: A single dose of placebo matched to trivalent influenza vaccine administered as intranasal spray on Day 1.
Period: Overall Study
Arm/Group | Trivalent Influenza Vaccine | Placebo
Started | 240 | 60 (One participant in this group received trivalent influenza vaccine on Day 1.)
Completed | 238 | 60
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trivalent Influenza Vaccine | Placebo | Total
Number analyzed (Participants) | 240 | 60 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (9.4) | 33.6 (9.0) | 33.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 34 | 171
  Male | 103 | 26 | 129

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Fever Greater Than or Equal to (>=) 101 Degrees Fahrenheit (F)
Description: Percentage of participants with fever defined as oral temperature >=101 degrees F were reported.
Time Frame: Within 7 days after vaccination
Population: Safety population included all participants who received any amount of investigational drug and had safety data available. Participants were included in the safety population according to the investigational drug received.
Measure: Number; unit: percentage of participants
Arm/Group | Trivalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 241 | 59
percentage of participants | 0.4 | 0.0
Statistical Analysis 1: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Non-Inferiority or Equivalence — Pre-specified equivalence criterion for fever within 7 days of vaccination mentioned that the upper limit of 95 percent (%) confidence interval (CI) for difference in percentage of participants with fever >=101 degrees F should be less than 5 percentage points; Percent difference = 0.4, 95% CI 2-sided [-5.3 to 2.6] — A two-sided 95% CI was constructed using the exact method based on the score statistic proposed by Chan and Zhang

2. Secondary Outcome: Percentage of Participants With Solicited Symptoms
Description: Solicited symptoms were predefined symptoms or events to be specifically inquired about and assessed daily after vaccine administration up to 14 days after vaccination. The solicited symptoms included fever greater than (>) 100.0 degrees F (37.8 degrees Celsius), runny nose, sore throat, cough, vomiting, muscle aches, chills, decreased activity and headache. Results are reported for all solicited symptoms except fever >=101 degrees F (reported as primary outcome) within 7 days after vaccination and all solicited symptoms within 14 days after vaccination.
Time Frame: Within 7 and 14 days after vaccination
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Trivalent Influenza Vaccine: A single dose of 10^(7.0 +/- 0.5) FFU of trivalent influenza vaccine administered as intranasal spray on Day 1.
Arm/Group | Trivalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 241 | 59
percentage of participants
  Any symptom within 7 days | 37.3 | 25.4
  Fever: greater than 100 degrees F within 7 days | 0.8 | 0.0
  Fever: greater than 102 degrees F within 7 days | 0.0 | 0.0
  Fever: greater than 103 degrees F within 7 days | 0.0 | 0.0
  Runny nose within 7 days | 20.7 | 11.9
  Sore throat within 7 days | 9.5 | 3.4
  Cough within 7 days | 4.6 | 5.1
  Vomiting within 7 days | 0.0 | 0.0
  Muscle aches within 7 days | 3.3 | 3.4
  Chills within 7 days | 1.7 | 0.0
  Decreased activity (tiredness) within 7 days | 10.0 | 6.8
  Headache within 7 days | 15.4 | 11.9
  Any symptom within 14 days | 39.4 | 27.1
  Fever: greater than 100 degrees F within 14 days | 1.2 | 0.0
  Fever: >= 101 degrees F within 14 days | 0.8 | 0.0
  Fever: greater than 102 degrees F within 14 days | 0.0 | 0.0
  Fever: greater than 103 degrees F within 14 days | 0.0 | 0.0
  Runny nose within 14 days | 21.6 | 11.9
  Sore throat within 14 days | 11.2 | 6.8
  Cough within 14 days | 5.4 | 5.1
  Vomiting within 14 days | 0.4 | 0.0
  Muscle aches within 14 days | 3.7 | 3.4
  Chills within 14 days | 2.5 | 0.0
  Decreased activity (tiredness) within 14 days | 11.2 | 6.8
  Headache within 14 days | 16.6 | 13.6
Statistical Analysis 1: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 11.9, 95% CI 2-sided [-1.9 to 23.9] — Any symptom within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 2: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.8, 95% CI 2-sided [-4.9 to 3.3] — Fever >100 degrees F within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 3: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-6.1 to 1.8] — Fever >102 degrees F within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 4: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-6.1 to 1.8] — Fever >103 degrees F within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 5: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 8.9, 95% CI 2-sided [-2.6 to 17.7] — Runny nose within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 6: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 6.2, 95% CI 2-sided [-2.2 to 11.6] — Sore throat within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 7: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = -0.5, 95% CI 2-sided [-9.3 to 4.7] — Cough within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 8: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-6.1 to 1.8] — Vomiting within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 9: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = -0.1, 95% CI 2-sided [-8.0 to 4.3] — Muscle aches within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 10: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 1.7, 95% CI 2-sided [-4.1 to 4.4] — Chills within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 11: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 3.2, 95% CI 2-sided [-6.5 to 9.8] — Decreased activity (tiredness) within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 12: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 3.5, 95% CI 2-sided [-7.8 to 11.9] — Headache within 7 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 13: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 12.3, 95% CI 2-sided [-1.6 to 24.4] — Any symptom within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 14: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 1.2, 95% CI 2-sided [-4.5 to 3.9] — Fever >100 degrees F within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 15: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.8, 95% CI 2-sided [-4.9 to 3.3] — Fever >=101 degrees F within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 16: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-6.1 to 1.8] — Fever >102 degrees F within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 17: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-6.1 to 1.8] — Fever >103 degrees F within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 18: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 9.7, 95% CI 2-sided [-1.8 to 18.6] — Runny nose within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 19: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 4.4, 95% CI 2-sided [-5.3 to 11.2] — Sore throat within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 20: Comparison: Trivalent Influenza Vaccine; Test type: Superiority or Other; Percent difference = 0.3, 95% CI 2-sided [-8.6 to 5.7] — Cough within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 21: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.4, 95% CI 2-sided [-5.3 to 2.6] — Vomiting within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 22: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 0.3, 95% CI 2-sided [-7.8 to 4.8] — Muscle aches within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 23: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 2.5, 95% CI 2-sided [-3.3 to 5.5] — Chills within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 24: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 4.4, 95% CI 2-sided [-5.3 to 11.2] — Decreased activity (tiredness) within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method
Statistical Analysis 25: Comparison: Trivalent Influenza Vaccine vs Placebo; Test type: Superiority or Other; Percent difference = 3.0, 95% CI 2-sided [-8.7 to 12.0] — Headache within 14 days of vaccination: Difference in percentage of participants and 95% CI were constructed based on Chan and Zhang's method

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs were events between administration of study drug and up to 14 days after vaccination that were absent before treatment or that worsened relative to pre-treatment state. Results are given for AEs reported within 7 days and 14 days after vaccination.
Time Frame: Within 7 and 14 days after vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 241 | 59
participants
  Within 7 days | 26 | 4
  Within 14 days | 28 | 5

4. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) and New Onset Chronic Diseases (NOCDs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent SAEs were serious events between administration of study drug and up to 180 days after the dose that were absent before treatment or that worsen relative to pretreatment state. An NOCD was a newly diagnosed medical condition that was of a chronic, ongoing nature and was assessed by the investigator as medically significant. Results are given for TESAEs and NOCDs reported within 28 days and 180 days after vaccination.
Time Frame: Within 28 and 180 days after vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 241 | 59
participants
  TESAEs within 28 days | 1 | 0
  TESAEs within 180 days | 1 | 2
  NOCDs within 28 days | 0 | 0
  NOCDs within 180 days | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Required Antipyretic and/or Analgesic Medication
Time Frame: Within 7 and 14 days after vaccination
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Trivalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 241 | 59
percentage of participants
  Anti-pyretic or analgesic within 7 days | 9.1 | 5.1
  Anti-pyretic and analgesic within 7 days | 8.7 | 5.1
  Anti-pyretic or analgesic within 14 days | 9.1 | 6.8
  Anti-pyretic and analgesic within 14 days | 8.7 | 6.8

ADVERSE EVENTS:
Time Frame: Serious Adverse events (SAEs): up to 180 days after vaccination; other adverse events (AEs): up to 14 days after vaccination
Description: Safety population included all participants who received any amount of investigational drug and had safety data available. Participants were included in the safety population according to the investigational drug received.
Groups:
- TRIVALENT VACCINE: A single dose of 10^(7.0 +/- 0.5) fluorescent focus units (FFU) of trivalent influenza vaccine administered as intranasal spray on Day 1.
Arm/Group | TRIVALENT VACCINE | PLACEBO
Serious Adverse Events (participants affected / at risk) | 1/241 | 2/59
Other Adverse Events (participants affected / at risk) | 28/241 | 5/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRIVALENT VACCINE (N=241) | PLACEBO (N=59)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRIVALENT VACCINE (N=241) | PLACEBO (N=59)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 3 (3)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.